CLINICAL TRIAL: NCT04856111
Title: A Study of the Efficacy and Safety of Pirfenidone vs. Nintedanib in the Treatment of Fibrotic Lung Disease After Coronavirus Disease-19 Pneumonia
Brief Title: Pirfenidone vs. Nintedanib for Fibrotic Lung Disease After Coronavirus Disease-19 Pneumonia
Acronym: PINCER
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Sahajal Dhooria, Assistant Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INT/IEC/2021/SPL-462
Record Dates: First submitted 2021-04-19; First posted 2021-04-22 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Novel Coronavirus-induced Lung Fibrosis
MeSH Terms: interventions — pirfenidone; nintedanib

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pirfenidone (Active Comparator): Pirfenidone will be started at a dose of 600 mg/day. The dose will be escalated by 600 mg/day every 3-7 days up to a targeted dose of 2400 mg/day. The subjects will be administered the maximum tolerated dose for a total period of 24 weeks from randomization.
  Interventions: Drug: Pirfenidone
- Nintedanib (Active Comparator): Subjects in this group will be administered nintedanib at a dose of 150 mg twice daily. The liver function tests will be monitored as above. The dose will be reduced to 100 mg twice daily, if there is intolerance to 300 mg/day dose.
  Interventions: Drug: Nintedanib

INTERVENTIONS:
Drug: Pirfenidone — Same as arm description
  Arms: Pirfenidone
Drug: Nintedanib — Same as arm description
  Arms: Nintedanib

SUMMARY:
The antifibrotic agents, namely pirfenidone and nintedanib have been found to be effective in the treatment of idiopathic pulmonary fibrosis (IPF). Nintedanib has also been found to be effective in treating systemic sclerosis-related interstitial lung disease (ILD) and non-IPF progressive fibrosing ILDs. Pirfenidone has also been found beneficial unclassifiable ILDs. Whether these drugs would be effective in treating post-COVID lung fibrosis also is unknown. As the final pathway of lung fibrosis appears to be common among different diffuse parenchymal lung diseases (DPLDs), it is hoped that these antifibrotic agents might be helpful in post-COVID fibrosis. There are no randomized studies that have assessed the role of pirfenidone or nintedanib in post COVID fibrosis. In the current study, we aim to assess the efficacy and safety of pirfenidone and compare it with nintedanib in the treatment of post-COVID lung fibrosis.

DETAILED DESCRIPTION:
Since the early part of 2020, the entire world has been affected by a pandemic of the coronavirus disease 2019 (COVID-19) caused by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). The disease has a short incubation period (median, 3 days) and is highly transmissible. This disease may manifest as an asymptomatic infection and through an entire range of symptoms of varying severity to severe, life-threatening disease. Although diverse systemic features might be present, the usual presentation is with lower respiratory tract involvement in the form of pneumonia often resulting in the development of the acute respiratory distress syndrome (ARDS). In some patients, multi-organ failure sets in, possibly as a result of a cytokine storm interplaying with a thrombotic microangiopathy.

Early lung disease is characterized pathologically by neutrophilic and exudative capillaritis in the lungs with some evidence of microthrombosis.2 This may be followed by a picture of diffuse alveolar damage along with ongoing intravascular thrombosis in the pulmonary vessels. In late stages, an organizing pneumonia (OP) develops with extensive proliferation of fibroblasts within the airspaces. Clinically, most patients make a complete recovery after COVID pneumonia. Other patients may demonstrate some signs of recovery from the acute illness with resolution of fever and recovery of organ functions, however they continue to have some degree of breathlessness, persistent infiltrates on radiologic studies, and/or hypoxemia. The CT abnormalities in these patients are commonly characterized by patchy, multifocal consolidation and ground-glass opacities suggestive of the OP pattern. Coarse reticulation and parenchymal bands may also be present.

Patients with such diffuse lung disease after COVID-19, herein referred to as post-COVID diffuse lung disease (PC-DLD) are often treated with glucocorticoids. Although most patients with a predominant OP pattern of injury would have a resolution of lung parenchymal abnormalities either spontaneously or with glucocorticoids, some of them might develop signs of lung fibrosis, in the form of traction bronchiectasis and/or honeycombing. Some subjects have ongoing respiratory symptoms despite treatment with steroids, and they may be found to have persistent reticulation or non-resolving consolidation on chest imaging that may represent early fibrosis.

The antifibrotic agents, namely pirfenidone and nintedanib have been found to be effective in the treatment of idiopathic pulmonary fibrosis (IPF). Nintedanib has also been found to be effective in treating systemic sclerosis-related interstitial lung disease (ILD) and non-IPF progressive fibrosing ILDs. Pirfenidone has also been found beneficial unclassifiable ILDs. Whether these drugs would be effective in treating post-COVID lung fibrosis also is unknown. As the final pathway of lung fibrosis appears to be common among different diffuse parenchymal lung diseases (DPLDs), it is hoped that these antifibrotic agents might be helpful in post-COVID fibrosis. There are no randomized studies that have assessed the role of pirfenidone or nintedanib in post COVID fibrosis. In the current study, we aim to assess the efficacy and safety of pirfenidone and compare it with nintedanib in the treatment of post-COVID lung fibrosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 years
2. Diagnosed to have COVID-19 by means of a real-time reverse transcription polymerase chain reaction (rRT-PCR) test performed on a respiratory (upper or lower respiratory) sample or positive IgM antibody test or a rapid antigen test with consistent clinicoradiologic findings within the previous 4 months
3. Persistent respiratory symptoms
4. Having post-COVID parenchymal involvement >10% of the lung parenchyma on visual inspection of the scans with the presence of radiologic signs of fibrosis (traction bronchiectasis/traction bronchiolectasis or honeycombing or reduced lung volumes), or having persistent reticulation or persistent consolidation despite a trial of glucocorticoids (minimum prednisolone dose of 10 mg/day, or equivalent) for a minimum period of 4 weeks after discharge for the acute COVID-19 illness

Exclusion Criteria:

1. Pregnant or lactating women
2. Having absolute contraindication for pirfenidone or nintedanib (advanced liver cirrhosis, persistent elevation of liver transaminases, documented hypersensitivity to pirfenidone or nintedanib, receiving anticoagulants or high dose aspirin or having a vascular stent in situ)
3. Known patient with diffuse lung disease prior to the diagnosis of COVID

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-03-17 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in the forced vital capacity (FVC) | 24 weeks
  Forced vital capacity will be measured using spirometry. The predicted value will be calculated based on standard reference equations.

SECONDARY OUTCOMES:
Proportion of subjects with improvement or stabilization | 24 weeks
  This will be defined by improvement or a <10% relative decline in FVC from the baseline value
Proportion of subjects with a good composite response | 24 weeks
  A good composite response will be defined as less than mMRC grade 2 breathlessness with ≥10% improvement in FVC with an oxygen saturation >92% during and after exertion.
Change in dyspnea score on modified Medical Research Council scale | 24 weeks
  The change in dyspnea score assessed using the modified Medical Research Council from the day of randomization to 6 weeks.The scale has a minimum score of 0 and a maximum score of 4, higher values indicate worse outcomes
Severity of dyspnea on the Functional Assessment of Chronic Illness Therapy - Dyspnea-10 item scale | 24 weeks
  Severity of dyspnea assessed using the Functional Assessment of Chronic Illness Therapy - Dyspnea-10 item scale. The scale has two item banks of 10 items each for dyspnea and functional limitations. EAch item has a minimum score of 0 and maximum score of 3. Higher scores represent worse outcomes.
Change in resting oxygen saturation | 24 weeks
  The change in resting oxygen saturation (measured by pulse oximetry) from the day of randomization to 24 weeks
Proportion of subjects with oxygen desaturation on exercise testing | 24 weeks
  Oxygen desaturation will be defined as a fall in oxygen saturation by 4% or more on exercise testing (by one-minute sit-to-stand test and six-minute walk test)
Percentage change in the six-minute walk distance | 24 weeks
  Six-minute walk test will be performed by trained technicians using a standard protocol
Proportion of participants who need rescue treatment | 24 weeks
  Rescue treatment would include the use of higher doses of glucocorticoids or other immunosuppressive agents
Change in health-related quality of life using the Short Form-36 questionnaire | 24 weeks
  Health-related quality of life assessed using Short Form-36 questionnaire. The questionnaire consists of 36 items covering 8 domains. Each domain score has a minimum value of 0 and maximum value of 100, with higher scores representing better outcomes
Change in respiratory health status using the King's Brief ILD questionnaire | 24 weeks
  Respiratory health status assessed using the King's Brief ILD questionnaire. The questionnaire has 15 items. The total score varies from 0 to 100, with higher scores representing better outcomes.
Changes in HRCT scores using the modified Salisbury system | 24 weeks
  Changes in HRCT scores for different features (reticulation, honeycombing, ground-glass opacities, mosaic attenuation/air trapping) will be calculated. The score for each feature range from 0 to 5 with higher scores representing worse outcomes
Proportion of subjects who develop adverse effects due to either study drug | 24 weeks
  The adverse effects of treatment (rash, hepatotoxicity, nausea, vomiting, diarrhea, headache, abdominal pain)
Predictors of response to antifibrotic agents, pirfenidone and nintedanib | 24 weeks
  These may include age, gender, the study group, baseline CT abnormalities, baseline FVC

CONTACTS AND LOCATIONS:
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No